CLINICAL TRIAL: NCT06891833
Title: A Randomized Controlled Phase II/III Clinical Study of BL-M07D1 With or Without Pertuzumab Versus Taxane + Trastuzumab and Pertuzumab in Neoadjuvant Therapy for HER2-Positive Breast Cancer
Brief Title: A Study of BL-M07D1 With or Without Pertuzumab Versus Taxane + Trastuzumab and Pertuzumab in Neoadjuvant Therapy for HER2-Positive Breast Cancer
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Sichuan Baili Pharmaceutical Co., Ltd. (Industry)
Collaborators: Baili-Bio (Chengdu) Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BL-M07D1-303
Record Dates: First submitted 2025-03-18; First posted 2025-03-24 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: HER2-positive Breast Cancer
MeSH Terms: interventions — pertuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study treatment (Experimental): Participants receive BL-M07D1 with or without Pertuzumab for the first cycle (3 weeks). Participants with clinical benefit could receive additional treatment for more cycles. The administration will be terminated because of disease progression or intolerable toxicity occurring or other reasons.
  Interventions: Drug: BL-M07D1; Drug: Pertuzumab

INTERVENTIONS:
Drug: BL-M07D1 — Administration by intravenous infusion for a cycle of 3 weeks.
Drug: Pertuzumab — Administration by intravenous infusion for a cycle of 3 weeks.

SUMMARY:
This trial is a registered phase III, randomized, open and multicenter study to evaluate the efficacy and safety of BL-M07D1 with or without Pertuzumab in the neoadjuvant treatment of HER2-positive breast cancer. The study is divided into a single-arm study phase (Phase II) and a randomized controlled study phase (Phase III).

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily signed informed consent and followed the program requirements;
2. Females ≥18 and ≤75 years of age at the time of signing the informed consent;
3. Expected survival time ≥6 months;
4. Patients with HER2-positive invasive breast cancer confirmed by histologic examination;
5. Clear hormone receptor (HR) status;
6. Clear clinical stage II-III based on American Joint Committee on Cancer (AJCC) staging 8th edition prior to neoadjuvant therapy;
7. Primary subjects without antitumor therapy for breast cancer;
8. Subjects consenting to mastectomy or breast-conserving surgery at the end of neoadjuvant therapy;
9. Radical surgery to the last dose of neoadjuvant therapy at least 2 weeks apart and up to 6 weeks apart;
10. Physical status score ECOG 0 or 1;
11. Organ function levels must be met provided that blood transfusions are not permitted within 14 days prior to the first administration of study drug, colony-stimulating factors are not permitted, and so on;
12. For premenopausal women of childbearing potential a pregnancy test must be performed within 7 days prior to initiation of treatment, serum pregnancy must be negative, and must be non-lactating; all enrolled patients should be using adequate and highly effective contraception throughout the treatment cycle and for 7 months after completion of treatment.

Exclusion Criteria:

1. Diagnosis of stage IV metastatic breast cancer;
2. Bilateral breast cancer;
3. Prior history of any breast cancer (unilateral or contralateral) other than lobular carcinoma in situ (LCIS);
4. Diagnosis of another primary malignancy within 5 years prior to first dose;
5. History of severe cardiovascular or cerebrovascular disease within 6 months prior to screening;
6. Prolonged QT interval, complete left bundle branch block, degree III atrioventricular block, and frequent and uncontrollable arrhythmias;
7. Poorly controlled hypertension (systolic blood pressure > 150 mmHg or diastolic blood pressure > 100 mmHg);
8. Complicated lung disease resulting in severely impaired lung function;
9. History of ILD / interstitial pneumonitis requiring steroid hormone therapy, current ILD / interstitial pneumonitis, or suspected of having such a disease, etc;
10. Human immunodeficiency virus antibody positivity, active hepatitis B virus infection, cirrhosis, or hepatitis C virus infection;
11. Severe infection within 4 weeks prior to first dose of study drug; active pulmonary inflammation present at screening;
12. Ongoing treatment with >10 mg/d prednisone systemic corticosteroid therapy or equivalent anti-inflammatory active drug or any form of immunosuppressive therapy within 2 weeks prior to the first dose;
13. Known hypersensitivity to the study therapeutic drug or any study drug excipients or other monoclonal antibodies;
14. Patients who are not suitable to receive the investigational drug (paclitaxel, patulizumab, trastuzumab);
15. Have a history of autologous or allogeneic stem cell transplantation or organ transplantation;
16. Suffering from severe neurological or psychiatric disorders;
17. Subjects with clinically significant bleeding or significant bleeding tendency within 4 weeks prior to signing the information;
18. Intestinal obstruction, Crohn's disease, ulcerative colitis or chronic diarrhea;
19. Subjects who are scheduled to receive a live vaccine or who have received a live vaccine within 28 days prior to the first dose;
20. Presence of other serious physical, laboratory test abnormalities or poor compliance that may increase the risk of participation in the study or interfere with the study results, as well as patients who, in the opinion of the investigator, are not suitable for participation in this study.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 120 (Estimated)
Dates: Start 2025-06-05 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Pathological complete response (pCR) rate | Up to approximately 48 months
  Pathological complete response (pCR) rate will be investigated.

SECONDARY OUTCOMES:
Event-free survival (EFS) | Up to approximately 48 months
  Event-free survival (EFS) is defined as the time between the day the subject is randomized and the first occurrence of any event.
Invasive disease-free survival (IDFS) | Up to approximately 48 months
  Invasive disease-free survival (IDFS) is defined as the time interval from the date of radical surgery to the presence of ipsilateral or contralateral recurrence of invasive breast cancer, locoregional recurrence, distant recurrence, or death from any cause, whichever occurs first.
Overall Survival (OS) | Up to approximately 48 months
  Overall survival (OS) is defined as the time between the day the subject is randomized and the subject's death.
Treatment Emergent Adverse Event (TEAE) | Up to approximately 48 months
  TEAE is defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally emerging, or any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a pre-existing condition during the treatment of BL-M07D1. The type, frequency and severity of TEAE will be evaluated during the treatment of BL-M07D1.

CONTACTS AND LOCATIONS:
Locations (30):
- China (30):
  - The First Affiliated Hospital of Bengbu Medical University, Bengbu, Anhui
  - Anhui Provincial Cancer Hospital, Hefei, Anhui
  - The First Affiliated Hospital of University of Science and Technology of China (Anhui Provincial Hospital), Hefei, Anhui
  - The First Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - Fujian Medical University Union Hospital, Fuzhou, Fujian
  - Guangdong Maternal and Child Health Center, Guangzhou, Guangdong
  - Sun Yat-Sen Memorial Hospital, Sun Yat-Sen University, Guangzhou, Guangdong
  - Cancer Hospital Chinese Academy of Medical Sciences, Shenzhen Center, Shenzhen, Guangdong
  - Liuzhou People's Hospital, Liuchow, Guangxi
  - Guangxi Medical University Cancer Hospital, Nanning, Guangxi
  - Hainan General Hospital, Haikou, Hainan
  - The Fourth Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - Xingtai People's Hospital, Xingtai, Hebei
  - Harbin Medical University Cancer Hospital, Harbin, Heilongjiang
  - Anyang Cancer Hospital, Anyang, Henan
  - The First Affiliated Hospital of Henan University of science and technology, Luoyang, Henan
  - Henan Provincial People's Hospital, Zhengzhou, Henan
  - Hunan Cancer Hospital, Changsha, Hunan
  - The Second Xiangya Hospital of Central South University, Changsha, Hunan
  - The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - Shaanxi Provincial People's Hospital, Xi'an, Shaanxi
  - The First Affiliated Hospital of Xi'an Jiaotong University, Xi'an, Shaanxi
  - Shandong Cancer Hospital, Jinan, Shandong
  - Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality
  - Shanxi Bethune Hospital, Taiyuan, Shanxi
  - Shanxi Cancer Hospital, Taiyuan, Shanxi
  - Sichuan Cancer Hospital, Chengdu, Sichuan
  - Tianjin Cancer Hospital, Tianjin, Tianjin Municipality
  - The First Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang